CLINICAL TRIAL: NCT02459873
Title: Modeling and Testing Change in Mental Abilities in Childhood Through Computer-based Interventions
Brief Title: Modeling and Testing Change in Mental Abilities in Childhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-01767
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Low Executive Function in Children

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer games to assess change in executive function skills (Experimental): Children in Intervention group get to train using executive function games at more difficult levels.
  Interventions: Behavioral: Computer games to assess change in executive function skills
- Easy games as active comparators for executive function skills (Active Comparator): Children in Non-intervention group get to play executive function games at an easy level.
  Interventions: Behavioral: Computer games to assess change in executive function skills

INTERVENTIONS:
Behavioral: Computer games to assess change in executive function skills — Children get access to computer games for 10 weeks for an hour each week.
  Other Names: Difficult / Easy games

SUMMARY:
Children with low executive function, working memory and attention skills in childhood not only do poorly at school, but also go on to do poorly on social, health, and financial indicators in adulthood.

The rate of executive function disorders in children is vastly underestimated at 17% , even when taking into account two of the more widely known disorders of Attention Deficit Hyperactivity Disorder (11%) and Fetal Alcohol Spectrum Disorders (6%), but children of lower socioeconomic status are especially vulnerable due to reduced resource availability.

As executive function, working memory and attention skills are central to success in later life, if children with low skills can be given targeted training to improve the skills they fall short on, there is potential to both improve their short-term academic performance, and influence long-term achievement. In fact, poor executive function skills and poor attention and working memory is a large predictor of poor performance even in typically developing children who are doing poorly academically.

Hypothesis 1. Those with lower working memory will also have lower problem solving skills and lower indices of other executive functioning skills such as reasoning/problem solving.

Hypothesis 2. Children that start with lower WM and PS will show the highest gains in training related performance, and such high gains on WM and PS will lead to better performance post-intervention compared to baseline measures of cognitive function.

Hypothesis 3: Those who make the largest gains in WM and PS with training will show more retention of training gains at 6 months compared those who show lower gains.

Aim 1. Assess working memory (WM) and processing speed (PS) skills in children and their inter-relationships with executive functioning skills Aim 2. Examine change in cognitive function in WM and PS after intensive training in WM and PS, during and immediately post-intervention Aim 3. Examine long-term retention of training effects on WM, PS, and executive functions.

The purpose of this study is to establish an effective and targeted working memory and processing speed intervention in children ages 7-10 with low to average executive function skills, by utilizing home-based computer games specifically designed to appeal to children.

Following institution approved consents, 60 low socioeconomic status children from Los Angeles will be recruited and enrolled in the study and be asked to play specific fun, but targeted cognitive computer games for 10 weeks.

The results of this pilot study will establish a protocol for feasibility of improving executive function skills in children with underdeveloped skills and inform on sufficiency of sample sizes, length of interventions, and directly impact computer-based intervention research and cost-effective techniques in children's cognitive development within the next 3-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Understands and speaks English

Exclusion Criteria:

* Diagnosed psychological disorder
* Head trauma with loss of consciousness of >5 minutes

Ages: 84 Months to 132 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Change in working memory skills assessed through Executive Function Battery and NIH ToolBox | 3 months
  Children will be assessed both on Executive Function Battery and the NIH Toolbox battery to examine change in working memory skills.
Change in processing speed skills assessed through Executive Function Battery and NIH ToolBox | 3 months
  Children will be assessed both on Executive Function Battery and the NIH Toolbox battery to examine change in processing speed skills.

SECONDARY OUTCOMES:
Change in school grades in science, reading and math. | 3-6 months
  Parents will be asked for children's school grades at the beginning of the study, during the study, and at the end of the study to assess the effects of the intervention
Change in parent reported behavior as assessed through BRIEF and CBCL questionnaires | 3-6 months
  Parental reports on BRIEF (Behavior Rating Inventory of Executive Function) and CBCL (Child Behavior Checklist) questionnaires will be used to assess change in behavior

CONTACTS AND LOCATIONS:
Overall Officials: Prapti Gautam, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States